CLINICAL TRIAL: NCT02303535
Title: National Congenital Heart Disease Audit
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: Society for Cardiothoracic Surgery in Great Britain & Ireland (Unknown); British Congenital Cardiac Association (Unknown)
Responsible Party: Sponsor
Other Study IDs: NICOR-CONGENITAL
Record Dates: First submitted 2014-11-25; First posted 2014-12-01 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-10

CONDITIONS: Congenital Heart Disease (CHD)
Keywords: Congenital heart disease; European Paediatric Cardiac Code Short List; Specific Procedure Definitions; OPCS; paediatric; pediatric
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Cardiac Surgical Procedures; Norwood Procedures; Heart Transplantation; Fontan Procedure; Arterial Switch Operation; Wound Healing; Surgical Procedures, Operative; Catheters; Radiofrequency Ablation; Defibrillators, Implantable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Congenital: All patients with congential and acquired heart disease treated by cardiac surgery and therapeutic cardiac catheterisations procedures .
  For acquired heart disease, the audit covers all arrhythmias & cardiomyopathies in patients less than 16 years old only.
  For congenital heart disease, the audit collects data on both children and adult patients.
  Interventions: Procedure: Cardiac Surgery; Procedure: Therapeutic cardiac catheterisations procedures

INTERVENTIONS:
Procedure: Cardiac Surgery — All patients with congential and acquired heart disease treated by cardiac surgery procedures.
  Other Names: Norwood procedure (Stage 1); Heart Transplant; TAPVD Repair + Arterial Shunt; Fontan procedure; Bidirectional cavopulmonary shunt; Senning or Mustard procedure; Truncus and interruption repair; Truncus arteriosus repair; Tricuspid valve replacement; Interrupted aortic arch repair; Multiple VSD Closure; Mitral valve replacement; Repair of total anomalous pulmonary venous drainage; Atrioventricular septal defect and tetralogy repair; Atrioventricular septal defect (complete) repair; Atrioventricular septal defect (partial) repair; Aortic valvotomy; Aortic valvoplasty; Anomalous coronary artery repair; Cor triatriatum repair; Arterial switch + VSD closure; Arterial switch (for isolated transposition); Pulmonary atresia VSD repair; Pulmonary valve replacement; Tetralogy with absent pulmonary valve repair; Tetralogy repair; Isolated coarctation repair; Aortic Valve Replacement - non Ross; Supravalvar aortic stenosis repair; Rastelli procedure; Aortic valve replacement - Ross; Aortic root replacement (not Ross); Subvalvar aortic stenosis repair; Aortopulmonary window repair; ASD repair; VSD Repair; Arterial shunt; Isolated Pulmonary artery band; PDA ligation (surgical)
Procedure: Therapeutic cardiac catheterisations procedures — All patients with congential and acquired heart disease treated by therapeutic cardiac catheterisations procedures .
  Other Names: Transcatheter PVR; VSD closure (catheter); Aortic balloon valvotomy; Coarctation angioplasty; Pulmonary artery stenting; ASD closure (catheter); PDA closure (catheter); Recoarctation angioplasty; Pulmonary balloon valvoplasty; Blade atrial septostomy; Coarctation stenting; PFO closure (catheter); Pulmonary valvotomy (radiofrequency); Duct Stenting; RVOT Stenting; Radiofrequency ablation for supraventricular tachycardia; Implantable Cardioverter Defibrillator

SUMMARY:
The National Institute of Cardiovascular Outcomes Research (NICOR) collects data and produces analysis to enable hospitals and healthcare improvement bodies to monitor and improve the quality of care and outcomes of cardiovascular patients.

The Congenital Heart Disease audit collects data on all cardiac surgery and therapeutic cardiac catheterisations procedures used to treat patients with congenital and acquired heart disease.

For acquired heart disease, the audit covers all arrhythmias & cardiomyopathies in patients less than 16 years old only. For congenital heart disease, the audit collects data on both children and adult patients. The audit covers all specialist centers in the UK and Republic of Ireland.

The project aims to improve the quality of care for children and adults with congenital heart disease by providing national comparative analysis of procedure specific activity and outcomes of cardiac surgery and therapeutic cardiac catheterisation procedures. The audit also provides quality indicators for the antenatal detection of major congenital heart disease.

The current dataset is available from here:

http://www.ucl.ac.uk/nicor/audits/congenital/datasets

DETAILED DESCRIPTION:
The Congenital Heart Disease audit collects data on all cardiac surgery and therapeutic cardiac catheterisations procedures used to treat patients with congenital and acquired heart disease

Data collection:

Hospitals use Patient Administration Systems and manual data entry by cardiac database managers to submit data to NICOR.

Data are either assimilated locally using third party commercial software and imported as a .csv file, or entered directly onto the NICOR database.

Data quality:

NICOR provide tools that communicate possible errors to centres submitting data. A data submitting schedule has been agreed with the centres, data is submitted and a validation report is returned each quarter. Centres are responsible for updating errors in the records.

An import log highlights missing and invalid data as well as records that failed to import due to data quality or compatibility issues.

In addition, data is validated by on site visits with a NICOR representative.

Data linkage:

Data is annually linked with Office fot National Statistics (ONS) life status and Hospital Episodes Statistics (HES) admission data to verify case ascertainment and to track long term outcome measures.

Information governance:

NICOR has Section 251 approval and data protection registration. An organisation-wide standard operating procedure is in place for Information Security Incident Management. University College London has a robust information governance framework, to which NICOR adheres.

ELIGIBILITY:
Inclusion Criteria:

Patient, judged by multidisciplinary team meeting as unsuitable for the procedure

Exclusion Criteria:

Patient, judged by multidisciplinary team meeting, as unsuitable for the procedure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All potential patients are assessed through a systematic process of clinical evaluation, diagnostic assessment. Patient selection is effected in each individual unit through a multidisciplinary team process. These teams consist not only of cardiac surgeons and interventional cardiologists but also of many other medical specialties and allied professionals. The decision as to the access route to be used is determined by the multidisciplinary team.
Sampling Method: Probability Sample
Enrollment: 120000 (Estimated)
Dates: Start 2000-04; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
30 day survival rates | 30 day survival from operation date
  The analysis shows the national survival rates at 30 days for each procedure and the national survival rates for individual procedures by age.

SECONDARY OUTCOMES:
1 year survival rates | 1 year survival rates after the date of the procedure
  Analysis include 1-year outcome but a death would not appear in the table until a full year has passed for the whole cohort of patients within that year. For example, the audit collection period is based on financial year of April 1st to March 31st. A patient that died in April would be reported within the same period as one that died 11 months later in March.

CONTACTS AND LOCATIONS:
Overall Officials: Rodney Franklin, MD, Study Chair — Royal Brompton & Harefield NHS Foundation Trust
Locations (10):
- United Kingdom (10):
  - Southampton General Hospital, Southampton, Hampshire
  - Royal Brompton Hospital, London, London
  - The Harley Street Clinic, London, London
  - Alder Hey Hospital, Liverpool, Merseyside
  - Royal Victoria Hospital Belfast, Belfast, Northern Ireland
  - John Radcliffe Hospital, Oxford, Oxfordshire
  - Freeman Hospital, Newcastle upon Tyne, Tyne and Wear
  - Leeds General Infirmary, Leeds, West Yorkshire
  - Queen Elizabeth Hospital (Edgbaston), Birmingham
  - The Heart Hospital, London

REFERENCES:
- [Background] Pagel C, Utley M, Crowe S, Witter T, Anderson D, Samson R, McLean A, Banks V, Tsang V, Brown K. Real time monitoring of risk-adjusted paediatric cardiac surgery outcomes using variable life-adjusted display: implementation in three UK centres. Heart. 2013 Oct;99(19):1445-50. doi: 10.1136/heartjnl-2013-303671. Epub 2013 Apr 5. PMID 23564473